CLINICAL TRIAL: NCT02524327
Title: Influence of the Modality of General Anesthesia Guided by the Bispectral Index (Manual or Automated) on the Occurrence of a Loss of Capability in Elderly Patients (> 70 Yrs): a Randomized Multicenter Study
Brief Title: Frail Status of Elderly Patients After Repair and Anesthesia Guided by the bispectraL Index
Acronym: FRAGIL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Material issues. Re-start in assessment
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2014/28; 2014-A01270-47 (Other: ANSM)
Record Dates: First submitted 2015-08-10; First posted 2015-08-14 (Estimated); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Anesthesia, General; Aged, 70 and Over
MeSH Terms: interventions — CDK13 protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Toolbox: Automated group (Experimental): Toolbox: Automated administration of intravenous anesthetic (propofol 1%) and analgesic (remifentanil, Ultiva(r)) guided by the Bispectral index through a controller with a previously described algorithm.
  Objective of depth anesthesia: 40-60
  Interventions: Other: Toolbox: Automated group
- Manual group (Active Comparator): Manual administration of intravenous anesthetic (propofol 1%) and analgesic (remifentanil, Ultiva(r)) guided by the Bispectral index as usually performed in the operative theater.
  Objective of depth anesthesia: 40-60
  Interventions: Other: Manual group

INTERVENTIONS:
Other: Toolbox: Automated group — A dedicated algorithm controls the infusion rate of drugs depending on the magnitude of variation of the bispectral index
  Other Names: controller
  Arms: Toolbox: Automated group
Other: Manual group — The anesthesiologist controls the infusion rate of drugs depending of the magnitude of variation of the bispectral index
  Arms: Manual group

SUMMARY:
The first aim of this study is to compare two methods of administration of intravenous anesthetics to obtain the same level of depth (bispectral index between 40 and 60): manual or automated and to determine a mid-term (6 months) influence of the frail phenotype on self-sufficient elderly patients after general anesthesia.

DETAILED DESCRIPTION:
To date, patients over the age of 60 yrs represent 25% of the population and are at increased risk of surgical repair. Reduction of postoperative morbidity and mortality are now two main concerns for medical research. Dependence on caregivers and cognitive impairments are two major risks in the elderly and even more in frail patients after surgery under general anesthesia. In this context continuous monitoring of the depth of anesthesia through bispectral index may reduce its occurrence with better control of too deep sedation periods (vasopressors…). Previous studies by the investigators' team suggest a better duration in the expected interval of Bispectral Index with automated control of administration of intravenous anesthetics guided by Bispectral Index. This method remains to be tested in this high-risk population. As a consequence, a randomization into two groups will be carried on elderly patients (> 70 yrs): manual administration of anesthetics guided by Bispectral Index (manual group) or automated administration (automated group). Complete preoperative assessments will determine the FRAIL status (with a decrease in the physiological reserve) and abilities of the patient according to the self-sufficient scale. At six months a follow-up will determine the geriatric status of the patient to explore the rate of impairment and to examine predictive factors in the preoperative assessment. Finally, the influence of the method of administration will be reported. Four hundred and thirty patients will be included in this multicenter study with 215 patients per group and stratification of the presence of a cancer and of the abdominal repair. The follow-up in this study allows the patient or his/her relatives to keep in touch with a physician and to prescribe some therapy early if frailty or any other cognitive impairment appears.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged > 70 years old
* American Society of Anesthesiologists class I to III
* Scheduled for abdominal surgery under total intra-venous anesthesia
* Self sufficient (living at home or in a non medical institution)
* Written consent to the study

Exclusion Criteria:

* Allergy to any intravenous agent (propofol or remifentanil)
* Cognitive impairment with a Mini Mental State Examination < 20
* Severe visual or hearing deficiency, apraxia
* Restriction of the use of bispectral index

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 134 (Actual)
Dates: Start 2015-07-07 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Rate of patients without occurrence of disability according to the InterRai scale | 6 months
  Disability is evaluated using the InterRai scale; a death is considered as an irreversible disability institutionalization is considered as a severe disability InterRai scale would discriminate other patients

SECONDARY OUTCOMES:
Mortality at day 28 | 28 days
Mortality at month 6 | 6 months
Rate of postoperative cognitive dysfunction | 6 months
  Cognitive dysfunction is evaluated using the Mini Mental State examination
Incidence of pneumopathy | 6 months
  Defined as a septic syndrome (fever) + increased number of polynuclear cells + typical image on chest X-ray + treatment with antibiotics
Incidence of pulmonary embolism | 6 months
  Diagnosis on CT-scan with contrast injection
Incidence of postoperative myocardial infarction | 6 months
  EKG modification and raised troponin
Incidence of evolution of the frail phenotype | 6 months
  Frail phenotype accordingly to Fried Scale
Quality of the general anesthesia | 1 day
  Defined as the time with a Bispectral Index in the interval 40-60
Performance of the automated system | 1 day
  Defined according to the Varvell score
Presence of Suppression Ratio | 1 day
  Defined as a period of isoelectric cortical signal with a threshold at 10% for 1 minute
Occurrence of arterial hypotension requiring treatment | 1 day
  Defined as a drop of 20% or more of the mean arterial pressure compared to the basal value measured before anesthetic induction and the requirement for a vasoactive agent
Patients'satisfaction about general anesthesia | 1 day
  Evaluation using a numeric scale from 0 (the worst remembrance) to 10 (an excellent moment)
Occurrence of awareness | 3 months
  Postoperative specific questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Morgan Le Guen, MD, Principal Investigator — Hopital Foch
Locations (4):
- France (4):
  - Hopital Jean Minjoz, Besançon
  - Institut Hopsitalier Franco-Britannique, Levallois-Perret
  - Centre Clinical, Soyaux
  - Hopital Foch, Suresnes

REFERENCES:
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Liu N, Chazot T, Hamada S, Landais A, Boichut N, Dussaussoy C, Trillat B, Beydon L, Samain E, Sessler DI, Fischler M. Closed-loop coadministration of propofol and remifentanil guided by bispectral index: a randomized multicenter study. Anesth Analg. 2011 Mar;112(3):546-57. doi: 10.1213/ANE.0b013e318205680b. Epub 2011 Jan 13. PMID 21233500
- [Derived] Le Guen M, Herr M, Bizard A, Bichon C, Boichut N, Chazot T, Liu N, Ankri J, Fischler M. Frailty Related to Anesthesia guided by the Index "bispectraL" (FRAIL) study: study protocol for a randomized controlled trial. Trials. 2017 Mar 16;18(1):127. doi: 10.1186/s13063-017-1868-9. PMID 28298244